CLINICAL TRIAL: NCT06773325
Title: The Effect of Buzzy Application on Pain and Comfort Level During Heel Blood Collection in Newborns: A Randomized Controlled Study
Brief Title: Buzzy Application During Heel Blood Collection in the Newborn
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Yuzuncu Yil University (Other)
Responsible Party: Principal Investigator, Veysel Can, Asst. Prof., Yuzuncu Yil University
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Health Services Research
Other Study IDs: Buzzy
Record Dates: First submitted 2025-01-02; First posted 2025-01-14 (Actual); Last update posted 2025-01-14 (Actual); Status verified 2025-01

CONDITIONS: Buzzy

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Buzzy (Experimental)
  Interventions: Behavioral: Buzzy application
- Control (No Intervention)

INTERVENTIONS:
Behavioral: Buzzy application — Buzzy application during heel prick blood collection
  Arms: Buzzy

SUMMARY:
Objective The aim of this study was to evaluate the effects of Buzzy device application during heel prick blood collection on pain level and comfort in newborns.

Method. The study was conducted in a Family Health Center affiliated to the Public Health Directorate of a province in eastern Turkey between September and November 2024 using a randomized controlled experimental design. The study sample consisted of 80 newborn infants born at 37-42 weeks gestational age and within the first 28 days of birth (Buzzy group: n = 40, control group: n = 40). The Buzzy group was treated by placing the Buzzy device approximately 30 seconds before heel prick blood collection. In the control group, routine heel prick was performed without any application. Neonatal introduction form, Neonatal Infant Pain Scale and Neonatal Comfort Behavior Scale were used for data collection.

ELIGIBILITY:
Inclusion Criteria:

* Those in the neonatal period between 0-28 days,
* voluntary participation of the parent,
* between 37-42 weeks of gestational age
* babies with vital signs within normal limits

Exclusion Criteria:

* The integrity of the skin in the area where the device was to be implanted was compromised,
* Nerve damage or deformity in the extremity to be heel bled,
* Genetic - with a congenital anomaly or congenital metabolic disorder,
* undergoing cardiopulmonary resuscitation,
* No heel prick on the first attempt,
* with osteogenesis imperfecta and infants given analgesics in the last 6 hours

Ages: 0 Days to 28 Days | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 80 (Actual)
Dates: Start 2024-09-01 (Actual); Primary Completion 2024-11-20 (Actual); Study Completion 2024-11-30 (Actual)

PRIMARY OUTCOMES:
The Neonatal Infant Pain Scale | pre-test post-test (approximately three months)
  min-max (0-7) , fewer points is a good result

CONTACTS AND LOCATIONS:
Locations (1):
- Van Yüzüncü Yıl University, Van, Tuşba, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No